CLINICAL TRIAL: NCT04036981
Title: The Effect of Muscle Selection for Botulinum Toxin A Injection on the Treatment Outcome in Poststroke Elbow Flexor Spasticity
Brief Title: Muscle Selection for Botulinum Toxin A Injection in Poststroke Elbow Flexor Spasticity
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ilker şengül, Principal Investigator, Izmir Katip Celebi University
Other Study IDs: 2018-KAE-0230
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Muscle Spasticity
Keywords: Stroke; Muscle spasticity; Botulinum toxin A
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Brachialis: Targeted muscle for BoNT A injection
  Interventions: Drug: Botulinum toxin type A
- Biceps: Targeted muscle for BoNT A injection
  Interventions: Drug: Botulinum toxin type A
- Brachialis plus Brachioradialis: Targeted muscles for BoNT A injection
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Injection of botulinum toxin A into the spastic elbow flexor muscle or muscles
  Other Names: Botox; Dysport

SUMMARY:
Botulinum toxin A (BoNT A) has been reported to be effective in the treatment of elbow flexor spasticity. Although BoNT A is an efficacious treatment option, there is a debate in the selection of target muscle(s) for BoNT injection in the treatment of poststroke elbow flexor spasticity. The decision of muscle selection for BoNT A injection is mostly made according to the physical examination findings in real life practice.One of the guiding findings in this decision is the position of the spastic arm.

In this study, hypothesis is that the change in severity of spasticity with BoNT A injection differs depending on the muscle selection in chronic stroke patients with elbow flexor and forearm pronator spasticity.

DETAILED DESCRIPTION:
Botulinum neurotoxin A (BoNT A) has been reported to be effective in the treatment of elbow flexor spasticity. In the treatment of poststroke elbow flexor spasticity with BoNT A, three main muscles injected individually or in combination are musculus biceps brachii, musculus brachialis and musculus brachioradialis. Although BoNT is an efficacious treatment option, there is a debate in the selection of target muscle(s) for BoNT A injection in the treatment of poststroke elbow flexor spasticity. Superficiality of the biceps brachii muscle makes it an easy target for botulinum toxin injection. In dynamic electromyography studies, it has been reported that brachioradialis muscle is the most common contributor one to elbow flexion spasticity, followed by biceps brachii muscle. In the diagnostic selective nerve blocks, the brachialis muscle has been reported to be foreground. In a recent study using the modified Delphi Method Design, the expert committee was only fully agree on the application of BoNT A into the brachioradialis muscle.

The decision of muscle selection for BoNT A injection is mostly made according to the physical examination findings in real life practice. One of the guiding findings in this decision is the position of the spastic arm. The typical pattern of spastic elbow and forearm in patients with stroke is characterized by flexion at the elbow, and pronation in the forearm. As far as the investigators know, there has not been carried out any study investigating the effect of muscle selection for BoNT application on the treatment outcome (severity of spasticity) in chronic stroke patients with elbow flexor and forearm pronator spasticity.

The aim of this study is to investigate whether treatment response (change in severity of spasticity) differs according to BoNT A injected muscle in chronic stroke patients with elbow flexor and forearm pronator spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Chronic (equal to or upper than 1 year) stroke patients with position of elbow flexion and forearm pronation while standing or sitting
* Grade 2 or 3 elbow flexor spasticity and grade 1 to 3 forearm pronator spasticity according to Modified Ashworth Scale
* Stage 2 or 3 Brunnstrom's motor recovery stage of upper extremity
* To agree to participate in the study

Exclusion Criteria:

* <18 years old
* Pregnancy
* Botulinum toxin injection within the last three months
* Presence of elbow contracture
* History of operation to spastic upper extremity
* Spasticity due to other causes other than stroke
* Do not agree to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke patients with elbow flexor and forearm pronator spasticity
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Dynamic Component of Spasticity (Spasticity Angle) | up to 4 week
  According to the Modified Tardieu Scale, the difference between the angle of slow passive motion and the angle of muscle reaction represents the dynamic component of spasticity (spasticity angle) in degree. A big difference suggests spasticity while the low difference suggests muscular contracture. In this study, dynamic component of spasticity (spasticity angle) of elbow joint at forearm pronation position will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Şengül, M.D., Principal Investigator — Izmir Katip Celebi University
Locations (1):
- İlker Şengül, Izmir, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keenan MA. Management of the spastic upper extremity in the neurologically impaired adult. Clin Orthop Relat Res. 1988 Aug;(233):116-25. PMID 3042230
- [Background] Genet F, Schnitzler A, Droz-Bartholet F, Salga M, Tatu L, Debaud C, Denormandie P, Parratte B. Successive motor nerve blocks to identify the muscles causing a spasticity pattern: example of the arm flexion pattern. J Anat. 2017 Jan;230(1):106-116. doi: 10.1111/joa.12538. Epub 2016 Sep 6. PMID 27595994
- [Background] Keenan MA, Haider TT, Stone LR. Dynamic electromyography to assess elbow spasticity. J Hand Surg Am. 1990 Jul;15(4):607-14. doi: 10.1016/s0363-5023(09)90023-5. PMID 2380525
- [Background] BASMAJIAN JV, LATIF A. Integrated actions and functions of the chief flexors of the elbow: a detailed electromyographic analysis. J Bone Joint Surg Am. 1957 Oct;39-A(5):1106-18. No abstract available. PMID 13475410
- [Background] Bohannon RW, Smith MB. Interrater reliability of a modified Ashworth scale of muscle spasticity. Phys Ther. 1987 Feb;67(2):206-7. doi: 10.1093/ptj/67.2.206. PMID 3809245
- [Background] Gracies JM, Bayle N, Vinti M, Alkandari S, Vu P, Loche CM, Colas C. Five-step clinical assessment in spastic paresis. Eur J Phys Rehabil Med. 2010 Sep;46(3):411-21. PMID 20927007
- [Background] Hefter H, Jost WH, Reissig A, Zakine B, Bakheit AM, Wissel J. Classification of posture in poststroke upper limb spasticity: a potential decision tool for botulinum toxin A treatment? Int J Rehabil Res. 2012 Sep;35(3):227-33. doi: 10.1097/MRR.0b013e328353e3d4. PMID 22555318
- [Background] Simpson DM, Patel AT, Alfaro A, Ayyoub Z, Charles D, Dashtipour K, Esquenazi A, Graham GD, McGuire JR, Odderson I. OnabotulinumtoxinA Injection for Poststroke Upper-Limb Spasticity: Guidance for Early Injectors From a Delphi Panel Process. PM R. 2017 Feb;9(2):136-148. doi: 10.1016/j.pmrj.2016.06.016. Epub 2016 Jun 23. PMID 27346090
- [Derived] Sengul I, Askin A, Tosun A. Effect of muscle selection for botulinum neurotoxin treatment on spasticity in patients with post-stroke elbow flexor muscle over-activity: an observational prospective study. Somatosens Mot Res. 2022 Mar;39(1):10-17. doi: 10.1080/08990220.2021.1986383. Epub 2021 Oct 10. PMID 34632927